CLINICAL TRIAL: NCT02636517
Title: Fecal Microbiome Transplant in Pediatric C. Difficile
Brief Title: Fecal Microbiome Transplant
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Judith Kelsen (Other)
Responsible Party: Sponsor-Investigator, Judith Kelsen, Attending Physician - CHCA, Children's Hospital of Philadelphia
Organization: Children's Hospital of Philadelphia (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-010531
Record Dates: First submitted 2015-12-16; First posted 2015-12-21 (Estimated); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Clostridium Difficile; Inflammatory Bowel Disease; Crohn's Disease; Ulcerative Colitis
Keywords: Fecal Microbiota transplant
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- C. Difficile without IBD (Other): Fecal Microbiota transplant in pediatric patients with recurrent C. Difficile
  Interventions: Biological: Fecal Microbiota Transplant
- C. Difficile with IBD (Other): Fecal Microbiota transplant in pediatric patients with recurrent C. Difficile with Inflammatory Bowel Disease
  Interventions: Biological: Fecal Microbiota Transplant

INTERVENTIONS:
Biological: Fecal Microbiota Transplant — Fecal Microbiota transplant via colonoscopy, considered both a biologic and a drug

SUMMARY:
Fecal Microbiota Transplant (FMT) in pediatric patients with recurrent C. Difficile with or without Inflammatory Bowel Disease (IBD)

The aims of this study are to determine the safety and efficacy of FMT treatment in pediatric patients with recurrent or moderate to severe C. Difficile without (through an observational study) and with (through a clinical trial) Inflammatory Bowel Disease and to determine the effect of FMT on the gut microbiota through the use of 454 pyrosequencing before and after transplantation in these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Inflammatory Bowel Disease by colonoscopy, radiographic and clinic measures, as per standard protocol.
2. Age ≥ 3 years old.
3. Recurrent C. difficile or Moderate to Severe C. difficile.
4. Satisfactory completion of the medical interview and physical exam conducted by a study team member
5. Participants must be between 3 and 21 years of age (inclusive)
6. Signed informed consent form, and assent (if applicable)

Exclusion Criteria:

1. Patients <3 years old
2. Patients with other co-morbid intestinal infectious processes
3. Recipients with a history of severe (anaphylactic) food allergy
4. If female, participants of childbearing potential (females aged 11 and older or those who have already begun menstruating) will be required to have a urine pregnancy test on the day of the FMT procedure. Patients who are pregnant will not be enrolled.
5. Patients with severe IBD.
6. Ongoing/anticipated antibiotic use for non-CDI indication
7. Adverse event attributable to a previous FMT
8. Patients with allergies to sodium chloride or glycerol, both ingredients Generally Recognized As Safe (GRAS)
9. Any other condition for which the treating physician thinks the treatment may pose a health risk
10. Predicted death within time period of follow-up
11. Patients who are on supraphysiologic doses of corticosteroids

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 250 (Estimated)
Dates: Start 2015-12; Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with a recurrence of C. difficile (CDI) | 7 days
  The hypothesis is that FMT will be an effective therapy for patients with IBD and CDI, resulting in resolution of symptoms as compared to historical controls on antibiotic therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Judith Kelsen, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No